CLINICAL TRIAL: NCT03419013
Title: A Pilot Evaluation of Newly Developed Adhesives and How They Are Impacted by Output
Brief Title: Evaluation of the Performance of an Adhesive Strip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP265_18
Record Dates: First submitted 2018-01-15; First posted 2018-02-01 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test of new adhesive strip (Experimental): A new adhesive strip has been developed and will be tested in this investigation
  Interventions: Other: New adhesive strip

INTERVENTIONS:
Other: New adhesive strip — This strip is made of a newly developed adhesive

SUMMARY:
This study investigated the performance of a new adhesive strip when impacted by output

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have had an ileostomy for more than one year
4. Have intact skin on the area used in the evaluation
5. Has an ileostomy with a diameter up to (≤) 35 mm
6. Have a peristomal area accessible for application of test product (assessed by investigator)

Exclusion Criteria:

1. Currently receiving or have within the past 2 month received radio- and/or chemotherapy
2. Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.
3. Are pregnant or breastfeeding
4. Having dermatological problems in the peristomal- or abdominal area (assessed by investigator)
5. Participating in other interventional clinical investigations or have previously participated in this investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Trans epidermal water loss | 24 hours
  trans epidermal water loss is a measure of the skins barrier function. There is always a oss of water from the skin due to evaporation. However, when the skin barrier is damaged this evaporation increases. Thus, trans epidermal water loss can be used to assess the skins barrier function

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Nielsen, Principal Investigator — Head of the pre-clinical department
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

IPD SHARING:
Plan to Share IPD: No